CLINICAL TRIAL: NCT03150173
Title: Buprenorphine Treatment at Syringe Exchanges to Reduce Opioid Misuse and HIV Risk
Brief Title: Onsite Buprenorphine Treatment at Syringe Exchange Programs
Acronym: O-BMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-7484; R01DA044878 (NIH)
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Opiate Addiction
Keywords: opioid use disorder, syringe exchange, HIV risk reduction
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to receive the O-BMT intervention or enhanced referral
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- O-BMT (onsite treatment) (Experimental): Over 2 weeks at the syringe-exchange program, participants in the O-BMT arm will see a buprenorphine provider twice, receive weekly blister packs of medication, and then their care will be transferred to a community health center for maintenance buprenorphine treatment
  Interventions: Behavioral: Onsite treatment; Drug: Buprenorphine
- Enhanced Referral (Active Comparator): In the control arm, participants will receive enhanced referral to a community health center for maintenance buprenorphine treatment
  Interventions: Behavioral: Enhanced referral; Drug: Buprenorphine

INTERVENTIONS:
Behavioral: Onsite treatment — Participants will see a buprenorphine treatment provider who will assess for clinical criteria for opioid use disorder and write a prescription for buprenorphine treatment, which will be filled in a community pharmacy.
  Arms: O-BMT (onsite treatment)
Behavioral: Enhanced referral — Participants will receive an expedited appointment at a community health center for evaluation for buprenorphine treatment
  Arms: Enhanced Referral
Drug: Buprenorphine — all participants will receive buprenorphine

SUMMARY:
This trial will recruit syringe exchange participants with opioid use disorder in New York City and test whether starting buprenorphine treatment at the syringe exchange program is more effective than referral to a community health center for buprenorphine treatment.

DETAILED DESCRIPTION:
In a 24 week randomized controlled trial based in a large urban area with high rates of opioid use disorder (OUD) and HIV, 250 out-of-treatment opioid users who utilize syringe exchanges will be recruited and randomize to receive an onsite treatment intervention (O-BMT) or enhanced referral to buprenorphine treatment. Over 2 weeks, participants in the O-BMT arm will see a buprenorphine provider twice, receive weekly blister packs of medication, and then their care will be transferred to a community health center for maintenance buprenorphine treatment. In the control arm, participants will receive enhanced referral to the community health center for maintenance buprenorphine treatment. Data collection will include urine drug tests, questionnaires, and medical and pharmacy record review. Key outcomes will include engagement in buprenorphine treatment, treatment outcomes, and programmatic costs. Buprenorphine diversion will be assessed by using electronic monitors that estimate medication adherence, testing urine samples for buprenorphine, and through sequential surveys regarding buying or selling illicit buprenorphine.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years
2. opioid use disorder
3. interest in buprenorphine treatment
4. motivation for opioid use disorder treatment
5. willingness to accept community health center referral
6. syringe exchange participant

Exclusion Criteria:

1. receiving opioid agonist treatment in the past 30 days (confirmed by New York Prescription Drug Monitoring Program);
2. inability to provide informed consent
3. unstable mental illness (e.g., suicidality, psychosis, etc.)
4. severe alcohol use disorder or benzodiazepine use disorder by the Diagnostic and Statistical Manual of Mental disorders, Fifth Edition (DSM-5) criteria
5. hypersensitivity to buprenorphine or naloxone.
6. pregnancy (confirmed via urine testing)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Fox, MD, MS, Principal Investigator — Associate Professor of Medicine
Locations (3):
- United States (3):
  - Washington Heights CORNER Project, New York, New York
  - New York Harm Reduction Educators, New York, New York
  - BOOM!Health Harm Reduction Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez-Correa A, Abbas B, Riback L, Ghiroli M, Norton B, Murphy S, Jakubowski A, Hayes BT, Cunningham CO, Fox AD. Onsite buprenorphine inductions at harm reduction agencies to increase treatment engagement and reduce HIV risk: Design and rationale. Contemp Clin Trials. 2022 Mar;114:106674. doi: 10.1016/j.cct.2021.106674. Epub 2022 Jan 3. PMID 34990854

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 211 participants were screened and 97 were randomized into the study. Of the 114 participants who were not enrolled into the study, 98 participants did not meet all of the eligibility criteria, 13 did not show up for the enrollment visit and 3 participants signed the informed consent form but were not randomized into the study.
Period: Overall Study
Arm/Group | O-BMT (Onsite Treatment) | Enhanced Referral
Started | 48 | 49
Completed | 35 | 44
Not Completed | 13 | 5
Not completed — Lost to Follow-up | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | O-BMT (Onsite Treatment) | Enhanced Referral | Total
Number analyzed (Participants) | 48 | 49 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (9.9) | 43.3 (11.3) | 42.0 (10.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 38 | 38 | 76
  Female | 9 | 10 | 19
  Transgender | 0 | 1 | 1
  Refuse to answer | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Black | 12 | 4 | 16
  Hispanic White | 5 | 4 | 9
  Hispanic Other | 13 | 14 | 27
  Non-Hispanic Black | 6 | 10 | 16
  Non-Hispanic White | 11 | 13 | 24
  Non-Hispanic Other | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 48 | 49 | 97
Mental Health Condition [Count of Participants; unit: Participants] — Mental health condition was assessed at baseline based on participant response to a survey question as to whether they have ever been diagnosed with a serious mental illness. The percentage of participants who responded "Yes" to having been diagnosed with a mental health condition is summarized by study arm.
  Participants | 22 | 22 | 44
Intravenous Drug Use [Count of Participants; unit: Participants] — Prior intravenous (IV) drug use was assessed at baseline by participant response to a dichotomous (Yes/No) query regarding previous IV drug use over the prior 30-day period. The percentage of participants who responded "Yes" to prior IV use is summarized by study arm.
  Participants | 28 | 33 | 61
Buprenorphine Use [Count of Participants; unit: Participants] — Prior Buprenorphine use was determined at baseline by participant response to a dichotomous (Yes/No) query regarding previous Buprenorphine usage in their lifetime. The percentage of participants who responded "Yes" to prior Buprenorphine use is summarized by study arm.
  Participants | 19 | 16 | 35
Opioid Use Disorder (OUD) Criteria [Mean (Standard Deviation); unit: criteria] — The mean number of OUD criteria (based on The American Psychiatric Association, Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, DSM-5, criteria) met per participant at baseline was summarized by study arm using basic descriptive statistics. The DSM-5 Checklist, an 11-item questionnaire measuring the number of diagnostic criteria for a substance use disorder met by an individual, has a range of 0-11 with a higher score representing more criteria met. The DSM-5 defines meeting 2-3 criteria as OUD mild, 4-5 criteria as OUD moderate, and 6 or more criteria as OUD severe.
  criteria | 10.5 (2.1) | 10.8 (2.2) | 10.7 (2.2)
Heroin use [Mean (Standard Deviation); unit: days] — The number of days of Heroin use over the prior 30-day period was assessed based on participant responses to a survey administered at baseline. Group mean values are summarized by study arm using basic descriptive statistics.
  days | 23.3 (11.3) | 24.2 (10.1) | 23.8 (10.7)
Methadone Use [Mean (Standard Deviation); unit: days] — The number of days of Methadone use over the prior 30-day period was assessed based on participant responses to a survey administered at baseline. Group mean values are summarized by study arm using basic descriptive statistics.
  days | 2.0 (7.3) | 0.6 (1.7) | 1.3 (4.5)
Opioid or Analgesic Use [Mean (Standard Deviation); unit: days] — The number of days of Opioid or Analgesic use over the prior 30-day period was assessed based on participant responses to a survey administered at baseline. Group mean values are summarized by study arm using basic descriptive statistics.
  days | 3.3 (8.5) | 3.3 (8.4) | 3.3 (8.4)
Alcohol Use [Mean (Standard Deviation); unit: days] — The number of days of Alcohol use over the prior 30-day period was assessed based on participant responses to a survey administered at baseline. Group mean values are summarized by study arm using basic descriptive statistics.
  days | 1.6 (4.9) | 1.3 (2.5) | 1.4 (3.7)
Cocaine Use [Mean (Standard Deviation); unit: days] — The number of days of Cocaine use over the prior 30-day period was assessed based on participant responses to a survey administered at baseline. Group mean values are summarized by study arm using basic descriptive statistics.
  days | 10.0 (11.4) | 12.6 (12.2) | 11.3 (11.8)
Amphetamine Use [Mean (Standard Deviation); unit: days] — The number of days of Amphetamine use over the prior 30-day period was assessed based on participant responses to a survey administered at baseline. Group mean values are summarized by study arm using basic descriptive statistics.
  days | 0.2 (0.8) | 0.9 (4.4) | 0.6 (2.7)
Polysubstance Use [Mean (Standard Deviation); unit: days] — The number of days of polysubstance use (i.e., 2 or more drugs taken together) over the prior 30-day period was assessed based on participant responses to a survey administered at baseline. Group mean values are summarized by study arm using basic descriptive statistics.
  days | 11.0 (12.3) | 12.0 (13.3) | 11.5 (12.8)

OUTCOME MEASURES:

1. Primary Outcome: Buprenorphine Engagement
Description: Buprenorphine engagement was defined as the number of participants having an active buprenorphine prescription at 30 days after randomization. Responses were tallied using a dichotomous (i.e., Yes/No) measure. Data are summarized by study arm.
Time Frame: 30 days after randomization
Population: Intention to treat (ITT) analysis design. All participants, including those who are lost to follow-up, are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | O-BMT (Onsite Treatment) | Enhanced Referral
Number analyzed (Participants) | 48 | 49
Participants | 19 | 19
Statistical Analysis 1: Comparison: O-BMT (Onsite Treatment) vs Enhanced Referral; Test type: Superiority; p = 0.94, Chi-squared

2. Secondary Outcome: Treatment Retention
Description: Treatment retention was assessed by the number/percentage of participants who had a medical visit AND active buprenorphine prescription each month after buprenorphine initiation for 6 months. Results are summarized by study arm.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | O-BMT (Onsite Treatment) | Enhanced Referral
Number analyzed (Participants) | 48 | 49
Participants | 2 | 6
Statistical Analysis 1: Comparison: O-BMT (Onsite Treatment) vs Enhanced Referral; Test type: Superiority; p = 0.148, Chi-squared

3. Secondary Outcome: HIV Risk Behaviors
Description: Change in HIV risk behaviors will be assessed using the HIV risk behavior survey. This survey, consisting of a dichotomous (yes/no) measure of injection risk, will be used based on self-report of at least one risk behavior (sharing syringes, not using bleach to clean syringes, sharing cookers, or front/back loading of syringes) reported during the interval. The number of participants demonstrating at least one risk behavior is during the 6 month interval is summarized by study arm.
Time Frame: 6 months
Population: HIV Risk behavior data was unable to be collected from 12 participants in the onsite buprenorphine treatment (O-BMT) study arm and 9 participants in the Enhanced referral study arm. Accordingly, there is no HIV risk behavior data to report for these participants.
Measure: Count of Participants; unit: Participants
Arm/Group | O-BMT (Onsite Treatment) | Enhanced Referral
Number analyzed (Participants) | 36 | 40
Participants | 5 | 4
Statistical Analysis 1: Comparison: O-BMT (Onsite Treatment) vs Enhanced Referral; Test type: Superiority; p = 0.6132, Regression, Logistic; Adjustment for baseline self-report of injection-related HIV risk behaviors in the past 30 days; Odds Ratio (OR) = 1.445, 95% CI 2-sided [0.347 to 6.018]

4. Secondary Outcome: Buprenorphine Diversion
Description: Buprenorphine diversion will be defined as having at least one problem behavior: non-adherence to prescribed medication on electronic monitoring, self-reported diversion, or a urine sample consistent with diversion during the 6 month interval. This outcome measure is used to determine how many participants sell or give away prescribed medication. The number of participants with at least one problem behavior is summarized by study arm.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | O-BMT (Onsite Treatment) | Enhanced Referral
Number analyzed (Participants) | 48 | 49
Participants | 8 | 2
Statistical Analysis 1: Comparison: O-BMT (Onsite Treatment) vs Enhanced Referral; Test type: Superiority; p = .051, Fisher Exact

5. Secondary Outcome: Incremental Cost-effectiveness Ratio (ICER)
Description: The ICER will be calculated by dividing the incremental mean cost of the O-BMT arm relative to the control arm by the incremental mean effectiveness of the O-BMT arm relative to the control arm. The primary economic effectiveness outcome will be the quality-adjusted life-year (QALY), a measure that incorporates both duration and health-related quality-of-life and is recommended as the primary economic effectiveness measure. ICER is a composite measure that incorporates QALYs (also reported as a separate outcome measure) and mean costs (also reported as a separate outcome measure).
Time Frame: 6 months
Measure: Number; unit: Ratio (US dollars/QALY)
Groups:
- O-BMT vs. Enhanced Referral: O-BMT intervention costs and effects on quality adjusted life years were compared to the costs and effects of enhanced referral for buprenorphine treatment.
Arm/Group | O-BMT vs. Enhanced Referral
Number analyzed (Participants) | 97
Ratio (US dollars/QALY) | -805067
Statistical Analysis 1: Comparison: O-BMT vs. Enhanced Referral; Test type: Superiority; probability of cost effectiveness = 0.94; Data generated from the bootstrapping process were used to construct cost-effectiveness acceptability curves (CEACs), which effectively measure the uncertainty around the ICER point estimate

6. Secondary Outcome: Quality-adjusted Life-years (QALYs) Gained
Description: The main economic effectiveness outcome will be the quality-adjusted life-year (QALY), a measure that incorporates both duration and health-related quality-of-life and is recommended as the primary economic effectiveness measure. Mean years gained are summarized by study arm.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: years gained
Arm/Group | O-BMT (Onsite Treatment) | Enhanced Referral
Number analyzed (Participants) | 48 | 49
years gained | 0.20 [0.18 to 0.21] | 0.17 [0.15 to 0.19]
Statistical Analysis 1: Comparison: O-BMT (Onsite Treatment) vs Enhanced Referral; Test type: Superiority; p = 0.10, non-parametric bootstrapping — This is an actual calculated value not a threshold value; Non-parametric bootstrapping of adjusted mean values with 1000 iterations

7. Secondary Outcome: Mean Difference in Total Costs
Description: Mean cost (in US dollars) of the O-BMT arm were compared to the control arm. The resource utilization and resulting cost of implementing and administering the O-BMT intervention were estimated using microcosting analysis and participant self-report. Mean costs (in US dollars) are summarized by study arm.
Time Frame: 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: US Dollars
Arm/Group | O-BMT (Onsite Treatment) | Enhanced Referral
Number analyzed (Participants) | 48 | 49
US Dollars | 2702.43 [1280.77 to 6825.75] | 26853.97 [7001.37 to 146995.55]
Statistical Analysis 1: Comparison: O-BMT (Onsite Treatment) vs Enhanced Referral; Test type: Superiority; p < 0.01, non-parametric bootstrapping — This is an actual calculated value not a threshold value; Non-parametric bootstrapping of adjusted mean values with 1000 iterations

8. Secondary Outcome: Time to First Buprenorphine Prescription
Description: Time to first buprenorphine prescription is defined as the amount of time, in days, from when a participant enrolled in the study to receipt of first buprenorphine prescription. Results are summarized by study arm using basic descriptive statistics.
Time Frame: 1 month
Population: Time to first buprenorphine prescription results data was only available, and reported, from the sub-group of participants that received a prescription.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | O-BMT (Onsite Treatment) | Enhanced Referral
Number analyzed (Participants) | 36 | 29
days | 3.0 (4.6) | 14.0 (20.9)
Statistical Analysis 1: Comparison: O-BMT (Onsite Treatment) vs Enhanced Referral; Test type: Superiority; p = 0.011, t-test, 2 sided

9. Secondary Outcome: Number/Percentage of Participants Who Received Any Buprenorphine Prescription
Description: The Number/percentage of participants who received any buprenorphine prescription is defined as the number/percentage of participants that filled at least one prescription for buprenorphine while enrolled in the study. Results are summarized by study arm.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | O-BMT (Onsite Treatment) | Enhanced Referral
Number analyzed (Participants) | 48 | 49
Participants | 36 | 29
Statistical Analysis 1: Comparison: O-BMT (Onsite Treatment) vs Enhanced Referral; Test type: Superiority; p = 0.098, Chi-squared

10. Secondary Outcome: Total Time Prescribed Buprenorphine
Description: Total time prescribed buprenorphine is defined as the amount of time in days that participants were prescribed buprenorphine during the study period. Results are summarized by study arm using basic descriptive statistics.
Time Frame: 6 months
Population: Total time prescribed buprenorphine results data was only available, and reported, from the sub-group of participants that received a prescription.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | O-BMT (Onsite Treatment) | Enhanced Referral
Number analyzed (Participants) | 36 | 29
days | 46.7 (32.9) | 56.6 (34.8)
Statistical Analysis 1: Comparison: O-BMT (Onsite Treatment) vs Enhanced Referral; Test type: Superiority; p = 0.256, t-test, 2 sided

11. Post Hoc Outcome: Buprenorphine Adherence (Self-reported)
Description: Buprenorphine Adherence (self-reported), defined as meeting the primary outcome of buprenorphine engagement and self-reporting buprenorphine use at 30 days, was assessed as a composite measure for sensitivity analysis. The number of participants who both maintained an active buprenorphine prescription at 30 days after randomization, based on a dichotomous (i.e., Yes/No) measure, AND self-reported having taken buprenorphine on 1 or more days during the 30-day period were tabulated. Data are summarized by study arm.
Time Frame: 30 days after randomization
Population: Self-reported buprenorphine use data was unable to be collected from 20 participants in the onsite buprenorphine treatment (O-BMT) study arm and 15 participants in the Enhanced referral study arm.
Measure: Count of Participants; unit: Participants
Arm/Group | O-BMT (Onsite Treatment) | Enhanced Referral
Number analyzed (Participants) | 28 | 34
Participants | 13 | 13

12. Post Hoc Outcome: Buprenorphine Adherence (Confirmed)
Description: Buprenorphine Adherence (confirmed) was defined as meeting the primary outcome and having a urine drug screen positive for buprenorphine at 30 days. This outcome was assessed as a composite measure for sensitivity analysis. The number of participants who both maintained an active buprenorphine prescription at 30 days after randomization, based on a dichotomous (i.e., Yes/No) measure, AND tested positive for Buprenorphine in their urine sample following the 30-day period were tabulated. Data are summarized by study arm.
Time Frame: 30 days after randomization
Population: Urine samples were unable to be collected from 26 participants in the onsite buprenorphine treatment (O-BMT) study arm and 23 participants in the Enhanced Referral study arm. As such, an assessment was unable to be made for these participants.
Measure: Count of Participants; unit: Participants
Arm/Group | O-BMT (Onsite Treatment) | Enhanced Referral
Number analyzed (Participants) | 22 | 26
Participants | 5 | 8

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | O-BMT (Onsite Treatment) | Enhanced Referral
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/48 | 2/49
Other Adverse Events (participants affected / at risk) | 2/48 | 1/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | O-BMT (Onsite Treatment) (N=48) | Enhanced Referral (N=49)
Opioid Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Pt overdosed on opioids while at syringe exchange program
Skin Infection (Abscess) (Infections and infestations) | 1 (1) | 0 (0) — Verbatim Term: Abscess - arm. Secondary to blood clot. Hospitalized for 3 days
Skin Infection (Methicillin-resistant Staphylococcus aureus) (Infections and infestations) | 0 (0) | 1 (1) — Verbatim term: Methicillin-resistant Staphylococcus aureus Infection. Hospitalized for 7 days
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | O-BMT (Onsite Treatment) (N=48) | Enhanced Referral (N=49)
Asthma Attack (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Transportation Accident (Injury, poisoning and procedural complications) | 0 | 1
Endometriosis pain (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT03150173/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT03150173/ICF_001.pdf